CLINICAL TRIAL: NCT03112525
Title: DAPHNE Study: Real-Life Observational Study to Evaluate the Impact of the CYP3A4/5/7 and P-gp Pharmacogenetics and Phenotypic Activity on the Pharmacokinetic Profile of the Direct Oral Anticoagulants Rivaroxaban and Apixaban in Hospitalised Patients
Brief Title: DAPHNE Study: Direct Anticoagulant PHarmacogeNEtic
Acronym: DAPHNE
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Victoria Rollason, Pharmacologist, University Hospital, Geneva
Other Study IDs: CCER 2016-01490
Record Dates: First submitted 2017-04-07; First posted 2017-04-13 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Anticoagulants and Bleeding Disorders
Keywords: rivaroxaban; apixaban; cytochrome; anticoagulant; transporter; polymorphism; genotyping; phenotyping
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient under Rivaroxaban
  Interventions: Diagnostic Test: CYP3A4/5 and P-gp phenotyping; Genetic: CYP3A4/5 and P-gp genotyping
- Patient under Apixaban
  Interventions: Diagnostic Test: CYP3A4/5 and P-gp phenotyping; Genetic: CYP3A4/5 and P-gp genotyping

INTERVENTIONS:
Diagnostic Test: CYP3A4/5 and P-gp phenotyping — Phenotyping using a simplified version of the Geneva cocktail
Genetic: CYP3A4/5 and P-gp genotyping — Selected CYP3A4, CYP3A5, CYP3A7 and ABCB1 single nucleotide polymorphism (SNP) determination

SUMMARY:
New/direct oral anticoagulants (NOAC/DOAC), like apixaban and rivaroxaban, are an interesting alternative to unfractionated or low molecular weight heparin relayed by oral anti-vitamin K anticoagulants (VKA) for the treatment of venous thromboembolism and atrial fibrillation. This new generation of anticoagulants directly inhibit a factor in the blood coagulation pathway and have a wide therapeutic range overcoming several practical issues associated with VKA therapy including the need of routine coagulation monitoring potentially simplifying patient management. However, despite this wide therapeutic range, a large interindividual dose variability related to factors such as age, body surface, smoking, concomitant diseases as well as differences in drug metabolism, could put susceptible patients at risk for uncontrolled bleeding. Both rivaroxaban and apixaban are cleared primarily via cytochrome P450 (CYP) mediated hepatic metabolism, mainly CYP3A, and renal excretion, involving the P-glycoprotein (P-gp). Both CYP3A and P-gp activity show important interindividual variations due to drug interactions and/or genetic polymorphisms in corresponding genes.

The aim of the current study is to evaluate the impact of cytochrome activity and relevant polymorphisms on rivaroxaban/apixaban dosage regimen or treatment efficacy in a hospital setting. The safety issue in this context is particularly relevant, since hospitalisation is linked to a modification of the patient's treatment with often an increase in the number of medications. The resulting changes in metabolism due to modified cytochrome and transporter activities could affect rivaroxaban/apixaban blood concentrations. Our central hypothesis is that genotype and/or phenotype in CYP3A4/5/7 or P-gp may influence the rivaroxaban/apixaban plasma concentration and increase the risk of thrombotic or hemorrhagic events. Thus, investigating how the patient's genotype and/or phenotype for CYP3A4/5/7 and P-gp could potentially alter the bio-disponibility of rivaroxaban and apixaban and therefore the risk to develop adverse events or inefficacy would be of particular interest.

ELIGIBILITY:
Inclusion Criteria:

* Understanding of French or English language and provide signed and dated informed consent form.
* Willing to comply with all study procedures and be available for the duration of the study.
* Male or female, aged 18 years or above.
* Diagnosed with atrial fibrillation, deep-vein thrombosis or pulmonary embolism and under rivaroxaban or apixaban drug treatment.

Exclusion Criteria:

* Participation in a clinical study that may interfere with participation in this study.
* Under rivaroxaban or apixaban for prophylaxis of deep-vein thrombosis and pulmonary embolism in patients undergoing knee or hip replacement surgery.
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.
* Known allergy to midazolam or to fexofenadine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation, pulmonary embolism or deep-vein thrombosis, treated or on long-term prophylaxis with rivaroxaban or apixaban in a real-life clinical setting. All patients will be recruited at the Geneva University Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-01-07 (Actual)

PRIMARY OUTCOMES:
Comparison Apixaban Area Under the Curve (AUC) according to patient CYP3A phenotype | 6 weeks
Comparison Rivaroxaban AUC according to patient P-gp phenotype | 6 weeks
Comparison Apixaban AUC according to patient CYP3A genotype | 6 weeks
Comparison Rivaroxaban AUC according to patient P-gp genotype | 6 weeks

SECONDARY OUTCOMES:
Comparison Apixaban AUC according to patient hepatic function | 6 weeks
Comparison Rivaroxaban AUC according to patient hepatic function | 6 weeks
Comparison Apixaban AUC according to patient renal function | 6 weeks
Comparison Rivaroxaban AUC according to patient renal function | 6 weeks
Comparison adverse event (bleeding) occurrence according to patient CYP3A phenotype | 6 weeks
Comparison adverse event (bleeding) occurrence according to patient P-gp phenotype | 6 weeks

OTHER OUTCOMES:
Comparison bleeding management outcomes | 6 weeks
  Recording of all interventions, procedures and outcomes related to any reported bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Jules Desmeules, Pr., Study Director — HUG; Victoria Rollason, Principal Investigator — HUG
Locations (1):
- HUG, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No